CLINICAL TRIAL: NCT05820178
Title: A Prospective Randomized Controlled Study of the Efficacy of tDCS and rTMS in Promoting Wakefulness in Patients With Early Disorders of Consciousness
Brief Title: tDCS and rTMS in Patients With Early Disorders of Consciousness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOC1
Record Dates: First submitted 2023-04-07; First posted 2023-04-19 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Disorder of Consciousness; Stroke; Ischemic-hypoxic Encephalopathy
Keywords: Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Consciousness Disorders; Stroke; Hypoxia-Ischemia, Brain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS treatment group (Experimental): On the basis of conventional treatment, tDCS was given on day 2 after enrollment for a total of 14 days, once a day.
  Interventions: Device: tDCS
- rTMS treatment group (Experimental): On the basis of conventional treatment, rTMS was given on day 2 after enrollment for a total of 14 days, once a day.
  Interventions: Device: rTMS
- conventional treatment group (No Intervention): Not receiving any neuromodulation treatment.

INTERVENTIONS:
Device: tDCS — On the basis of conventional treatment, tDCS was given on day 2 after enrollment for a total of 14 days, once a day.
  Arms: tDCS treatment group
Device: rTMS — On the basis of conventional treatment, rTMS was given on day 2 after enrollment for a total of 14 days, once a day.
  Arms: rTMS treatment group

SUMMARY:
A randomized controlled study was conducted to explore the efficacy of early transcranial direct current stimulation (tDCS) and repetitive transcranial magnetic stimulation (rTMS) to promote wakefulness in patients with disorder of consciousness (DOC). In order to improve the prognosis of DOC patients with nontraumatic brain injury, we compared the effects of tDCS and rTMS on clinical behavior and neurophysiological performance, and selected a wake-up technique that could improve the prognosis of DOC patients with nontraumatic brain injury as early as possible, so as to reduce the pain of patients and their loved ones, and to reduce the economic burden of society and families.

DETAILED DESCRIPTION:
To study the efficacy of wakefulness promotion in patients with acute DOC due to severe non-traumatic brain injury (including stroke and ischemic-hypoxic encephalopathy), patients with early DOC were randomly divided into conventional treatment group, tDCS treatment group and rTMS treatment group for 14 consecutive days. Clinical scoring, evoked potential assessment, resting-state high-density electroencephalogram(EEG) and TMS-EEG assessment with functional analysis of brain network connectivity were applied for multidimensional assessment of brain function before and after wake-up promotion treatment (day 1 and day 15 of enrollment) to explore non-invasive brain stimulation(NIBS) techniques that can be performed at the bedside - tDCS, rTMS intervention The prognostic follow-up was performed at 3 months, 6 months and 12 months after DOC to compare the awakening rate after tDCS and rTMS prolongation treatment, and to preferably select an effective prolongation technique for early DOC. The safety of tDCS and rTMS was also clarified by comparing the differences in adverse effects and complications between tDCS treatment group and rTMS treatment group and conventional treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years
2. diagnosis of stroke or ischemic-hypoxic encephalopathy confirmed by neuroimaging (head MRI)
3. DOC, Glasgow coma score (GCS) <12 4.2-4 weeks of DOC

5.informed consent obtained from the patient's legal representative.

Exclusion Criteria:

1. foreign bodies such as metal or electronic devices in the skull (inside or on the surface of the tissue at the treatment stimulation site)
2. pacemaker or cochlear implants
3. history of epilepsy and family history of epilepsy
4. large cranial defects
5. significant cerebral edema lesions in both DLPFC
6. pregnant women
7. with severe physical diseases such as heart, lung, liver and kidney
8. brain death
9. new intracerebral lesions in patients during the study period affecting the assessment and prognosis, e.g. new stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
CRS-R | day 15 of enrollment
  The unabbreviated scale title is the coma recovery scale-revised.The CRS-R tests six components: auditory, language, visual, communication, motor and arousal levels, with a total score of 0-23. The lower the score, the more severe the brain damage and the deeper the DOC level.

SECONDARY OUTCOMES:
GCS | day 15 of enrollment
  The unabbreviated scale title is Glasgow coma score. The GCS tested 3 components: eye opening response, verbal response and motor response, with a total score of 15. The lower the score, the more severe the brain damage and the deeper the degree of DOC.
FOUR | day 15 of enrollment
  The unabbreviated scale title is full outline of unresponsiveness. The FOUR tested 4 components: eye opening response, brainstem reflex, respiratory pattern and motor response, with a total score of 0-16. The lower the score, the more severe the brain damage and the deeper the degree of DOC.
MMN | day 15 of enrollment
  The unabbreviated scale title is mismatch negative, representing an important component of auditory event-related potentials. We measure the occurrence, latency and wave amplitude of MMN.
MEP | day 15 of enrollment
  The unabbreviated scale title is motor evoked potential, which can examine the overall synchronization and integrity of the motor nerve transmission and conduction pathways from the cortex to the muscle. We measure the occurrence, latency and wave amplitude of MEP.
ABCD model of neural oscillation | day 15 of enrollment
  The total frequency content of the EEG is represented by a power spectrum that indicates the neural oscillations at different frequencies within the EEG signal. the ABCD model roughly classifies these changes in the EEG power spectrum into four types of ABCD, and this model is thought to reflect the severity of thalamo-cortical neural afferent block and is used to understand the different degrees of structural and functional afferent impairment present in patients with DOC. The ABCD model can reflect neural oscillations from A to D corresponding to the level of consciousness from DOC to wakefulness.
brain network transfer entropy | day 15 of enrollment
  Information flow between neural networks is the basis for understanding brain signal processing and function. Using the method of transfer entropy to analyze the information flow between two two channels, the wavelet consistency algorithm was applied to reveal the linear and nonlinear correlations between regional local field potentials, and the real-time coupling relationship between two channels of neural signals in time-frequency space, including coupling strength and coupling direction. Brain network connectivity can be determined, and comatose patients have significantly weaker connectivity than normal whole brain.
brain network phase synchronization | day 15 of enrollment
  The synchronization relationship between two two channels was analyzed using the method of phase synchronization to form a whole-brain synchronization matrix, and the synchronization matrix was calculated to analyze the direction and strength of whole-brain network connectivity by analyzing data such as shortest path and agglomeration coefficient in the small-world network index. Brain network connectivity can be determined, and comatose patients have significantly weaker connectivity than normal whole brain.
Prognostic scores (mRS) | 3 months, 6 months, 12 months after DOC
  The unabbreviated scale title is modified Rankin Scale. The mRS includes 0-6, and the higher the score, the worse the prognosis.
Prognostic scores (GOS) | 3 months, 6 months, 12 months after DOC
  The unabbreviated scale title is Glasgow Outcome Scale. GOS includes a score of 1-5, with the higher the score, the better the prognosis.
Prognostic scores (CRS-R) | 3 months, 6 months, 12 months after DOC
  The unabbreviated scale title is the coma recovery scale-revised. The CRS-R includes a total score of 0-23.The lower the score, the worse the prognosis.

IPD SHARING:
Plan to Share IPD: Yes
study protocol can be shared.
Supporting Information: Study Protocol
Time Frame: after Dec 2023, always
Access Criteria: email to authors